CLINICAL TRIAL: NCT02177734
Title: An Observer-blind Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Influenza Vaccine(s) GSK3277510A and GSK3277509A Administered in Adults 18 to 60 Years of Age
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Influenza Vaccine(s) GSK3277510A and GSK3277509A in Adults 18 to 60 Years of Age
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was cancelled for scientifically legitimate reasons not related to safety or efficacy of the vaccine.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201300; 2014-000796-27 (EudraCT Number)
Record Dates: First submitted 2014-06-19; First posted 2014-06-30 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Influenza
Keywords: Adjuvant; Safety; Influenza; H7N9; Immunogenicity; Adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Formulation 1 Group (Experimental): Subjects in this group will receive two doses of GSK3277510A H7N9 vaccine formulation 1 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3277510A
- Formulation 2 Group (Experimental): Subjects in this group will receive two doses of GSK3277510A H7N9 vaccine formulation 2 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3277510A
- Formulation 3 Group (Experimental): Subjects in this group will receive two doses of GSK3277510A H7N9 vaccine formulation 3 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3277510A
- Formulation 4 Group (Experimental): Subjects in this group will receive two doses of GSK3277510A H7N9 vaccine formulation 4 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3277510A
- Formulation 5 Group (Experimental): Subjects in this group will receive two doses of GSK3277509A H7N9 vaccine formulation 5 at a 21 day interval
  Interventions: Biological: Investigational H7N9 vaccine GSK3277509A
- Placebo Group (Placebo Comparator): Subjects in this group will receive two doses of placebo at a 21 day interval
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Investigational H7N9 vaccine GSK3277510A — One dose of GSK3277510A H7N9 vaccine administered intramuscularly (IM) in the deltoid region of non-dominant arm at Day 0 and the second dose of GSK3277510A H7N9 vaccine administered IM in the deltoid region of dominant arm at Day 21
  Arms: Formulation 1 Group; Formulation 2 Group; Formulation 3 Group; Formulation 4 Group
Biological: Investigational H7N9 vaccine GSK3277509A — One dose of GSK3277509A H7N9 vaccine administered IM at the deltoid region of non-dominant arm at Day 0 and the second dose of GSK3277509A H7N9 vaccine administered IM at the deltoid region of dominant arm at Day 21
  Arms: Formulation 5 Group
Biological: Placebo — One dose of placebo administered IM at the deltoid region of non-dominant arm at Day 0 and the second dose of placebo administered IM at the deltoid region of dominant arm at Day 21
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of different formulations of GSK Biologicals' H7N9 influenza vaccine in subjects 18 to 60 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults who are 18 to 60years of age (inclusive) at the time of first study vaccination.
* Written informed consent obtained from subject.
* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Healthy subjects as established by medical history and physical examination.
* Access to a consistent means of telephone contact.
* For subjects who undergo a screening visit: Results of screening safety laboratory tests that figure in eligibility assessment must be within reference ranges before dosing.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if they

  * have practiced adequate contraception for 30 days prior to vaccination, and
  * have a negative pregnancy test on the day of vaccination, and agree to continue to practice adequate contraception until 2 months after the last dose administered.

Exclusion Criteria:

* Presence or evidence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence or evidence of substance abuse.
* Diagnosed with cancer, or treatment for cancer within three years.
* Diagnosed with excessive daytime sleepiness, or narcolepsy; or history of narcolepsy in a subject's parent, sibling or child.
* Presence of a temperature ≥ 38.0ºC (≥100.4ºF), or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids within 30 days prior to the first dose of study vaccine/placebo, or any other cytotoxic, immunosuppressive or immune-modifying drugs within 6 months of first study vaccine/ placebo dose.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin.
* An acute evolving neurological disorder or Guillain Barré Syndrome within 42 days of receipt of prior seasonal or pandemic influenza vaccine.
* Administration of an inactive vaccine within 14 days or of a live attenuated vaccine within 30 days before the first dose of study vaccine/placebo.
* Planned administration of any vaccine other than the study vaccine/placebo before blood sampling at the Day 42 visit.
* Previous administration of any H7 vaccine or physician-confirmed H7 disease.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine/placebo, or planned use during the study period.
* Receipt of any immunoglobulins and/or any blood products within 90 days before the first dose of study vaccine/placebo, or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine including a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result before the first dose of study vaccine/placebo.
* Lactating or nursing women.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Humoral immune response in terms of vaccine-homologous hemagglutination inhibition (HI) antibody titers | At Day 42.
Occurrence of each solicited local symptom | During a 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after each vaccination.
Occurrence of each solicited general symptom | During a 7-day follow-up period (i.e., day of vaccination and 6 subsequent days) after each vaccination.
Occurrence of clinical safety laboratory abnormalities reported for samples | At the Day 0, 7, 21, 28 and 42 visits.
Occurrence of unsolicited adverse events (AEs) | 21 days after each dose.
Occurrence of Medically Attended Adverse Events (MAEs), potential Immune Mediated Diseases (pIMDs) and Serious Adverse Events (SAEs)[Active Phase] | From Day 0 until Day 42.

SECONDARY OUTCOMES:
Evaluation of adjuvant effect as assessed by vaccine-homologous hemagglutination inhibition (HI) antibody titers | At Day 42.
Humoral immune response in terms of vaccine-homologous hemagglutination inhibition (HI) antibody titers for plain antigen vaccine group | At Day 42.
Humoral immune response in terms of vaccine-homologous (H7N9) HI antibody titers. | GMTs and Seropositivity rates at Days 0, 21, 42 and Months 6 and 12. SCR and MGI at Days 21, 42 (Placebo group only) and Months 6 and 12. SPR at Days 0, 21, 42 (Placebo group only) and Months 6 and 12.
Humoral immune response in terms of vaccine-homologous (H7N9) neutralizing (MN) antibody titres. | GMTs and Seropositivity rates at the Days 0, 21, 42 and Month 6 visits. VRR at Days 21, 42 and Month 6 visits.
Humoral immune response in terms of vaccine-homologous (H7N9) HI antibody titers by age stratum. | GMTs, Seropositivity rates and SPR at Days 0, 21, 42 and Months 6 and 12. SCR and MGI at Days 21, 42 and Months 6 and 12.
Humoral immune response in terms of vaccine homologous (H7N9) neutralizing (MN) antibody titers for each study group by age stratum (18-40 years; 41-60 years) | GMTs and Seropositivity rates at Days 0, 21, 42 and Month 6. VRR at Days 21, 42 and Month 6.
Occurrence of MAEs, pIMDs and SAEs | Until the Month 12 visit.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline